



#### **CONSENT FORM**

Study Title: Effects of Nystatin Topical Oral Application on Oral Microbial Community

Principal Investigator: Jin Xiao, DDS, PhD

This consent form describes a research study, what you may expect if you decide to take part and important information to help you make your decision. Please read this form carefully and ask questions about anything that is not clear before you agree to participate. You may take this consent form home to think about and discuss with family or friends.

#### **Key Information**

- Being in this research study is voluntary it is your choice.
- You are being asked to take part in this study because you are a healthy adult and
  willing to help us find out whether a prescription oral rinse will affect the composition
  of bacteria and yeast in the mouth. A sample from your saliva will be collected to
  determine whether you are eligible to participate in this study depending on the
  amount of bacteria and yeast in your mouth.
- The purpose of this study is to find out whether a prescription oral rinse (Nystatin) application can reduce the number of bacteria and yeast in your mouth.
- Your participation in this study will last about three months and include 4 visits. Each visit may take approximately 15 to 30 minutes.
- Procedures will include:
  - o saliva (spit) and dental plaque sample collection
  - o filling out a questionnaire about your brushing, eating habits and other dental activities
  - o a complete dental exam
  - o rinsing your mouth with the prescription mouth rinse
  - o document in a daily diary that you have used the prescribed mouth rinse usage

RSRB Case Number: 0004638 

Version Date: 7/18/2020

- Your electronic medical/dental record will be accessed to review your medical history.
- There are risks from participating.
  - o The most serious risk is allergic reaction to study medication (Nystatin)
  - o The most common risk is loss of confidentiality
  - Other serious risks are side effects, including vomiting, nausea, diarrhea, and abdominal pain. See the "Risks of Participation" section in this consent form for more information. You should discuss these risks in detail with the study team.
- You cannot take part in this study if:
  - you are currently pregnant or breastfeeding, or you are planning to become pregnant during the next 3 months
  - you have a known allergy to Nystatin oral rinse
- You will not benefit from being in this study.
- You do not need to take part in this study, if you do not want to, it is your choice. Not
  participating will not affect your care received at Eastman Institute for Oral Health
  (EIOH).

### **Purpose of Study**

The purpose of this study is to find out whether a prescription oral rinse (Nystatin) application can reduce the number of bacteria and yeast in your mouth. A sample from your saliva will be collected to determine whether you are eligible to participate in this study depending on the amount of bacteria and yeast in your mouth. However, having a the amount of yeast in your mouth that makes you eligible for this study doesn't necessarily mean that you have a medical condition requiring a treatment. Results from this study may help us understand the effect that Nystatin oral rinse may have on certain type of oral bacteria, which may also cause tooth decay.

#### **Description of Study Procedures**

If you decide to take part in this study, you will be asked to attend four visits. The following study procedures will be completed:

#### Screening Visit/Enrollment (length of visit: Approximately 20 minutes)

The goal of the screening visit is to learn if you are eligible to take part in the remainder of the study. You may be eligible to take part in the study if: you have a certain level of oral yeast and bacteria in your mouth, you do not have any health conditions that would prevent you from using the study drug (Nystatin), and you are not currently breastfeeding, pregnant or planning to become pregnant within the next three months. The following activities will take place at the screening visit.

RSRB Case Number: 0004638 

Version Date: 07/18/2020

- a. If you are a patient of record at Eastman Institute for Oral Health, we will review your electronic medical/dental record to review your medical history. If you are not a patient of record, we will ask you to self-report medical background. We will conduct a free dental examination for you. If you have clinical diagnosis of oral candidiasis you be referred immediately for treatment.
- b. If you meet the initial eligibility for this study based on the dental exam and your medical history, we will invite you to participate.
- c. Once you agree to participate in this, and sign the consent form, we will collect a saliva (spit) sample if you had nothing to not eat, drink or did not brush your teeth within the past 2 hours. We will collect approximately 2 mL (less than ½ a teaspoon) of your saliva (spit) to screen for presence of oral yeast and bacteria that can cause a tooth decay. If you have brushed your teeth and had something to eat and drink within the past 2 hours, we will give you a choice to wait until the 2 hours requirement or reschedule this screening appointment.
- d. We will process your saliva sample and will inform you of the results within 3 days (72 hours). According to the results you may and may not be eligible to participate in the study depending on the amount of candida in your saliva. If you are eligible to participate in the study, this doesn't mean that you have a disease that require treatment.
- e. If you are eligible for the study we will schedule the first visit.
- f. A pregnancy test (urine test) will be conducted (if female).

# <u>Visit 1 (Day 0) (Approximately 2 weeks after screening visit) (length of visit: Approximately 30 minutes)</u>

- a) Comprehensive oral examination will be conducted such as checking your teeth, gums and other areas in your mouth.
- b) We will collect a saliva sample.
- c) We will collect plague around your gum lines.
- d) You will be asked to complete a questionnaire regarding your brushing, eating and other daily activities.
- e) We will give you a 1-week supply of Nystatin mouth rinse with the instructions for rinsing for two minutes, followed by spitting out the suspension four times a day (every four hours) for 1 week. Do not eat or drink anything for 30 minutes after using nystatin oral suspension in order to increase contact time with the mouth surface.
- f) We will also give you a diary to document Nystatin usage.

## Visit 2 (Approximately day 8-14) (Immediately after oral rinse visit) (length of

RSRB Case Number: 0004638 


## visit: Approximately 15 minutes)

- a) We will collect the unused remainder of the Nystatin bottle and diary.
- b) We will collect the saliva and plaque samples. These will be used to measure the amount of bacteria and yeast in your mouth.

## <u>Visit 3 (Approximately day 70-110) (3-month post oral rinse visit) (length of visit: Approximately 15 minutes)</u>

- c) We will collect saliva and plaque samples. These will be used to measure the amount of bacteria and yeast in your mouth.
- Information about your study participation and study results may be included in your electronic health record. If you have concerns about this or to obtain more detail, you should discuss this with the study team.
- If coming to the EIOH clinic is not convenient to you, you have the option to complete study visits at your home. With your permission, two study investigators will complete study visits at your home. The researchers are required to report information regarding potential child abuse or neglect reported by you or observed by them at your home during the research visit. The researcher will also report if there is a reasonable suspicion, based on information provided by you or observed during the research visit at your home, that you may present a danger of harm to others or that you may harm yourself unless protective measures are taken.
- With your permission, we will send you text messages to remind you about your upcoming study visit. The text message will include the location and time of your visit. We will not include your name in the text messages to protect your confidentiality. There might be cost for the text messages you receive from our study team. If you do not want to receive text messages at any time during the study period, please notify our study team, and we will not send the text messages to you.

#### **Number of Subjects**

Approximately 100 subjects will take part in this study at the Eastman Institute for Oral Health at the University of Rochester.

#### **Risks of Participation**

There are risks associated with using Nystatin. If you experience any of life threatening side effects, such as an allergic reaction discontinue its use and report to emergency department or call 911 immediately, and then inform study team. If you have any other

RSRB Case Number: 0004638 


concerns, please call the study investigator's phone number (585) 273-1957 and below are possible side effects:

- Bitter taste and stomach problems, including vomiting, nausea, diarrhea, and abdominal pain (most common).
- Rash, itching, fast heartbeat, breathing problems, facial swelling and muscle aches (rarely reported). This could be related to an allergic reaction to Nystatin.
- Overdose could cause nausea and stomach upset.

If you are a female of childbearing age who is pregnant, planning to become pregnant within the next three months, or if you are currently breastfeeding, you cannot take part in this study. If you learn that you are pregnant during the week that you are using Nystatin, you should consult your primary care physician and inform us.

As with any study, there is a possibility of breach of confidentiality. Appropriate precautions will be taken and procedures will be followed to maintain your confidentiality. To minimize this risk we will assign you a unique study number instead of your name or other personal information we collect about you. Information will be stored in a secure manner accessible to study personnel only. As you complete the questionnaire, you may skip a question if you do not want to answer. In addition, there may be a minor discomfort as we collect a bacteria sample around your gums. We will take the necessary precaution to minimize any discomfort.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this website at any time.

The study team may be notified if you receive other health care services at URMC or its Affiliates (e.g., visit to the emergency room). In addition, the following individuals may know you participated in research and may see results of testing conducted for this study:

- Staff at the University of Rochester Medical Center and its Affiliates (e.g., Strong Memorial Hospital, Highland Hospital, URMC primary care, specialist physician offices) who have a reason to access your electronic health record.
- Health care providers who are involved in your care at a facility that is not part of the University of Rochester Medical Center and its Affiliates and who have reason to access your electronic health record.
- Individuals who request a copy of information from your health record for activities such as treatment or payment (e.g., medical insurance companies, worker's compensation)

RSRB Case Number: 0004638 


## **Benefits of Participation**

The possible direct benefits may include the early detection of dental problems. If dental problems are identified you should follow up with your dentist for further treatment. If you do not have an established dentist, we will refer you to the URMC Eastman Institute for Oral Health clinic. Subjects will be informed that they/their health insurance provider will be responsible for any cost associated with treatment for any clinical conditions (other than Candida) that are identified.

#### **Compensation for Injury**

If you are directly injured by the Nystatin medication being studied, or by medical procedures needed because of this study, and you receive medical care for the injury, you may need to pay for that care. You will be reimbursed for reasonable and necessary medical costs for such care, but you might not be reimbursed for care covered and paid for by a third party like your health insurance provider, or costs such as required co-payments or deductibles related to that coverage. No other funds have been set aside to pay for such things as lost wages or expenses due to a current underlying illness or condition.

If your research injury is paid for by the University of Rochester, we will collect your name, date of birth, gender, and Medicare Health Insurance Claim Number or Social Security Number to determine your Medicare status. This information will be used only in accordance with the law. If you are a Medicare beneficiary, information about the study you are in, and any payments made related to your injury, will be reported to the Centers for Medicare & Medicaid Services (CMS), in accordance with CMS requirements. This information will not be used for any other purpose.

#### Costs

There will be no cost to you to participate in this study. However, your health insurance provider will be responsible for any cost associated with treatment for any clinical conditions (other than Candida) that are identified.

#### **Payments**

You and/or your insurance company will not be billed for any procedures done for the research. You could receive up to a total of \$50 gift cards for taking part in this study. You will receive \$10 gift card upon the completion of each of initial screening visit, first visit and second visit, and an additional \$20 gift card upon the completion of the last study visit for a total of \$50 in the form of gift cards. You will be provided with a parking voucher for each study visit you attend.

RSRB Case Number: 0004638 


## <u>Confidentiality of Records and Authorization to Use and Disclose Information for</u> Research Purposes

The University of Rochester makes every effort to keep the information collected from you private. In order to do so, we will assign a study number. Your study information, identified only by this study number, will be kept in a secure, locked cabinet in a secure room. All electronic files will be kept on a password protected computer in a secure, locked office. Sometimes, however, researchers need to share information that may identify you with people that work for the University, regulators or the study sponsor.

If you have never received a copy of the University of Rochester Medical Center (URMC) and Affiliates Notice of Privacy Practices, please ask the investigator for one.

What information may be used and given to others?

The study doctor will get your personal and medical information. For example:

- Research records
- Records about phone calls made as part of this research
- Records about your study visits
- Past and present medical records related to the study, including records of external providers that are available via your electronic health record at URMC & Affiliates
- Results of medical tests

Who may use and give out information about you?

- The study doctor and the study staff
- URMC and Affiliates

Your information may be given to:

- The Department of Health and Human Services
- The University of Rochester
- The Food and Drug Administration

Why will this information be used and/or given to others?

- To do the research
- To study the results
- To see if the research was done correctly

If the results of this study are made public, information that identifies you will not be used.

What if I decide not to give permission to use and give out my health information? Then you will not be able to be in this research study.

RSRB Case Number: 0004638 


May I review or copy my information? Yes, but only after the research is over.

How long will this permission be valid? This permission will last indefinitely.

May I cancel my permission to use and disclose information?

Yes. You may cancel your permission to use and disclose your health information at any time. You do this by sending written notice to the study doctor. Upon receiving the written notice, the study team will no longer use or disclose your health information and you will not be able to stay in this study. Information that has already been gathered may need to be used and given to others for the validity of the study.

#### May I withdraw from the study?

Yes. If you withdraw your permission to be in the study, no new health information identifying you will be gathered after that date. Information that has already been gathered may still be used and given to others.

Is my health information protected after it has been given to others?

No. There is a risk that your information will be given to others without your permission.

## Future Use of Information/Samples

Your information collected as part of this research will not be distributed or used for future research studies.

#### **Circumstances for Dismissal**

You may be withdrawn from the study if you do not keep appointments for study visits or if you cannot complete study activities.

### **New Study Information**

You may be withdrawn from the study if you do not keep appointments for study visits or if you cannot complete study activities.

#### **Contact Persons**

For more information concerning this research or if you feel that your participation has resulted in any research related injury, emotional or physical discomfort, please contact: Dr. Jin Xiao at (585) 273-1957

Please contact the University of Rochester Research Subjects Review Board at 265 Crittenden Blvd., CU 420628, Rochester, NY 14642, Telephone (585) 276-0005 or (877) 449-4441 for the following reasons:

RSRB Case Number: 0004638 


- You wish to talk to someone other than the research staff about your rights as a research subject;
- To voice concerns about the research;
- To provide input concerning the research process;
- In the event the study staff could not be reached.

## **Voluntary Participation**

Taking part in this study is voluntary. You are free not to take part or to withdraw at any time, for whatever reason. No matter what decision you make, there will be no penalty or loss of benefit to which you are entitled. In the event that you do withdraw from this study, the information you have already provided will be kept in a confidential manner.

This will not affect your class standing or grades. You will not be offered or receive any special consideration if you take part in this research.

Taking part in this research is not a part of your duties, and refusing will not affect your job. You will not be offered or receive any special job-related consideration if you take part in this research.

\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*


RSRB Case Number: 0004638 Version Date: 07/18/2020

RSRB Approval Date: 1/12/2021

Expiration Date: 1/11/2022

## **SIGNATURES/DATES**

After reading and discussing the information in this consent form you should understand:

- · Why this study is being done;
- · What will happen during the study;
- Any possible risks and benefits to you;
- Other options you may have instead of being in the study;
- How your personal information will be protected;
- What to do if you have problems or questions about this study.

| Text messaging opt in/out | | | |
|---|---|---|---|
| ☐ Yes, you may send text messaging to my phone. | | | |
| □ No, you may not send text messaging to my phone. □ No, I do not have a phone Subject Consent I have read (or have had read to me) the contents of this consent form and have been encouraged to ask questions. I have received answers to my questions. I agree to participate in this study. I have received (or will receive) a signed copy of this form for my records and future reference. | | | |
| | | Subject Name (Printed by Subject) | |
| | | Signature of Subject | Date |
| Person Obtaining Consent | | | |
| I have read this form to the subject and/or the subject has r | ead this form. I will provide | | |
| the subject with a signed copy of this consent form. An exp | | | |
| given and questions from the subject were solicited and an | | | |
| satisfaction. In my judgment, the subject has demonstrated information. I have given the subject adequate opportunity signing. | | | |
| Name and Title (Print) | | | |
| Signature of Person Obtaining Consent | Date | | |